CLINICAL TRIAL: NCT04081363
Title: A Pilot Phase 2a, Multicenter, Open-label, Single-dose Trial to Assess the Pharmacokinetics of Centanafadine Extended-release Capsules After Oral Administration in Pediatric Subjects (9 to 12 Years, Inclusive) With Attention-deficit Hyperactivity Disorder
Brief Title: Open-label, Single-dose Trial to Assess the Pharmacokinetics of Centanafadine Extended-release Capsules in Pediatric Participants With Attention-deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 405-201-00037
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Intervention Model Description: All the participants received only centanafadine but divided into 2 arm groups based on administration (as capsules or drug sprinkled onto applesauce).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Swallowed Capsules Cohort (Experimental): Participants swallowed two capsules of centanafadine (one containing a 50-milligram [mg] dose as extended release beads and other containing a 5-mg dose as immediate-release [IR] beads), total dose of 55 mg, orally in the morning of Day 1 following a minimum 8-hour fast.
  Interventions: Drug: Centanafadine
- Sprinkled Onto Applesauce Cohort (Experimental): Participants were administered centanafadine 55 mg, contents of 2 capsules (one containing a 50-mg dose as beads and other containing a 5-mg dose as IR beads) sprinkled on a tablespoon of applesauce, orally in the morning of Day 1 following a minimum 8-hour fast.
  Interventions: Drug: Centanafadine

INTERVENTIONS:
Drug: Centanafadine — Extended-release and immediate-release capsules.
  Other Names: EB-1020

SUMMARY:
With the pharmacokinetics (PK) of centanafadine currently being evaluated in adults. The PK of extended-release centanafadine may differ in children compared to adults due to physiological differences in the gastrointestinal tract. The information in this trial will support pediatric dose selection in future trials.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from a legally acceptable representative and assent obtained from the participant prior to the initiation of any trial-related procedures.
* Male or female participants 9 to 12 years of age, inclusive, at the time of informed consent.
* Participants with documented history of ADHD and confirmation of an ADHD prescription medication.
* Participant is judged by the investigator to be clinically stable and has not had any psychiatric hospitalizations within the past 12 weeks.

Exclusion Criteria:

* Participants with a history of intellectual disability as determined by at least 1 of the following: intelligence quotient (IQ) < 70, or clinical evidence, or a social or school history that is suggestive of an intellectual disability.
* Participants who have any of the following:

  * Significant risk of committing suicide based on history
  * Current suicidal behavior
  * Imminent risk of injury to self
  * Active suicidal ideation
  * Any lifetime history of suicidal behavior detected by the "Baseline/Screening" version of the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Participants with a lifetime history of a substance use disorder (as determined by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition [DSM-5] criteria), or current substance misuse including alcohol and benzodiazepines, but excluding caffeine and nicotine.
* Participants with hypothyroidism or hyperthyroidism or an abnormal result for free thyroxine (T4) at screening.
* Participants who currently have clinically significant neurological, dermatological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders.
* Participants with insulin-dependent diabetes mellitus.
* Participants with epilepsy or a history of seizures or a history of severe head trauma or cerebrovascular disease.
* Any major surgery within 30 days prior to dosing with the investigational medicinal product (IMP).
* Any history of significant bleeding or hemorrhagic tendencies.
* Blood transfusion within 30 days prior to dosing with IMP.
* Participants with a positive drug screen for cocaine, marijuana (even if by prescription), or other illicit drugs, or alcohol, are excluded and may not be retested or rescreened.
* Participants who have a supine or standing diastolic blood pressure, after resting for at least 5 minutes ≥ 95 mmHg.
* Participants who participated in a clinical trial and were exposed to IMP within the last 30 days prior to screening or who participated in more than 2 interventional clinical trials within the past year.
* Participants with a history of true allergic response to a medication or a history of dermatologic adverse reactions or anaphylaxis secondary to drug exposure.
* Participants who do not tolerate venipuncture or have poor venous access that would cause difficulty when collecting blood samples.
* Relatives of the trial site employees cannot participate in the trial.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 07 October 2019 to 21 December 2019.
Pre-assignment Details: A total of 20 participants were screened and 13 participants were enrolled in the study to receive centanafadine as capsules or sprinkled onto applesauce.
Period: Overall Study
Arm/Group | Swallowed Capsules Cohort | Sprinkled Onto Applesauce Cohort
Started | 7 | 6
Completed | 6 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled analysis set included all participants who had eligibility to enroll in the trial based on screening process.
Groups:
- Total: Total of all reporting groups
Arm/Group | Swallowed Capsules Cohort | Sprinkled Onto Applesauce Cohort | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (1.0) | 10.5 (1.4) | 10.5 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: Maximum Plasma Concentration (Cmax) of Centanafadine
Time Frame: 1, 2, 3, 4, 6, 8, 10,12 hours post dose on Day 1 and 22-26 hours post dose on Day 2
Population: Pharmacokinetic (PK) analysis set included all participants who received the single dose of centanafadine and had at least 1 postdose evaluable plasma concentration.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Swallowed Capsules Cohort | Sprinkled Onto Applesauce Cohort
Number analyzed (Participants) | 6 | 6
nanograms per milliliter (ng/mL) | 153 (51.4) | 129 (52.8)

2. Primary Outcome: PK Parameter: Time to Maximum Plasma Concentration (Tmax) of Centanafadine
Time Frame: 1, 2, 3, 4, 6, 8, 10,12 hours post dose on Day 1 and 22-26 hours post dose on Day 2
Population: PK analysis set included all participants who received the single dose of centanafadine and had at least 1 postdose evaluable plasma concentration.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Swallowed Capsules Cohort | Sprinkled Onto Applesauce Cohort
Number analyzed (Participants) | 6 | 6
hours (h) | 3.03 [2.00 to 10.00] | 2.58 [1.03 to 6.00]

3. Primary Outcome: PK Parameter: Area Under Concentration-time Curve From Time 0 to 12 Hours Postdose (AUC0-12h) of Centanafadine
Time Frame: 0 to 12 hours post dose on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Swallowed Capsules Cohort | Sprinkled Onto Applesauce Cohort
Number analyzed (Participants) | 6 | 6
h*ng/mL | 962 (320) | 828 (346)

ADVERSE EVENTS:
Time Frame: Screening up to last follow-up (approximately 30 days)
Description: Safety analysis set included all participants who received the single dose of centanafadine.
Arm/Group | Swallowed Capsules Cohort | Sprinkled Onto Applesauce Cohort
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 1/7 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Swallowed Capsules Cohort (N=7) | Sprinkled Onto Applesauce Cohort (N=6)
Vessel Puncture Site Bruise (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT04081363/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT04081363/SAP_001.pdf